CLINICAL TRIAL: NCT02750150
Title: A Randomized Trial to Evaluate Freezed-dried Plasma in the Initial Management of Coagulopathy in Trauma Patients
Brief Title: Freeze-dried Plasma in the Initial Management of Coagulopathy in Trauma Patients
Acronym: TrauCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011_61; 2012-A00075-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-04-05; First posted 2016-04-25 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2016-04

CONDITIONS: Trauma; Coagulopathy
MeSH Terms: conditions — Wounds and Injuries; Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Freezed-dried plasma (Experimental): transfusion of 4 units of freezed dried plasma when available in patients at risk pf massive bleeding (transfusion of 4 red blood cells units in the first 6 hours after trauma)
  Interventions: Drug: Freezed-dried plasma
- Fresh-frozen plasma (Active Comparator): transfusion of 4 units of fresh frozen plasma when available in patients at risk pf massive bleeding (transfusion of 4 red blood cells units in the first 6 hours after trauma)
  Interventions: Drug: Fresh-frozen plasma

INTERVENTIONS:
Drug: Freezed-dried plasma — early transfusion of 4 units of freezed dried plasma
  Arms: Freezed-dried plasma
Drug: Fresh-frozen plasma
  Arms: Fresh-frozen plasma

SUMMARY:
Knowledge and management of bleeding in severe trauma has changed. A specific coagulopathy is present in 40% of cases. It has a very early onset and this coagulopathy is associated with increased mortality. It must be detected and treated early, as illustrated by the military medical data, from the Iraq war and civilian medicine. However, fresh frozen plasma (FFP) requires a thawing step.The French army has encouraged the development of a freeze-dried plasma of innovative because viral inactivation and universal blood grouping, well tolerated, with a reduced risk of TRALI. This sophisticated therapeutic product can be administered after 6 minutes of reconstitution without the need for cross-matching. Nevertheless, its used is currently reserved for military purpose in overseas operations and needs to be evaluated for civil use. To this end, the investigators need to evaluate the impact on coagulopathy of an immediate availability of plasma.

ELIGIBILITY:
Inclusion Criteria:

* Emergency
* Trauma patient admitted in participating trauma care centers
* Severe bleeding requiring transfusion with 4 units of red blood cells and 4 emergency plasma.
* Inclusion performed within the first 6 hours after trauma.

Exclusion Criteria:

* Patient taking anticoagulants
* Patients who have received hemostatic treatment during transport (tranexamic -acid excluded)
* Minor Patient
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-07-09 (Actual); Primary Completion 2016-04-17 (Actual); Study Completion 2016-04-17 (Actual)

PRIMARY OUTCOMES:
fibrinogen concentration (clauss) | 45 minutes after the admission on day 1 after trauma

SECONDARY OUTCOMES:
time frame of transfusion of 4 plasma | time range between the intention to transfuse plasma and the end of transfusion of 4 plasma within the first 6 hours after admission

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Susen, MD,PhD, Study Chair — University Hospital, Lille
Locations (1):
- Emergency unit, Salengro hospital,, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided